CLINICAL TRIAL: NCT00078312
Title: A 12-Month, Open-Label, Flexible-Dosage (100 to 250 mg/Day) Study of the Safety and Efficacy of CEP-10953 in the Treatment of Patients With Excessive Sleepiness Associated With Narcolepsy, Obstructive Sleep Apnea/Hypopnea Syndrome, or Chronic Shift Work Sleep Disorder (With an Open-Ended Extension Period)
Brief Title: Armodafinil (CEP-10953) for Treatment of Narcolepsy, Obstructive Sleep Apnea/Hypopnea Syndrome, or Chronic Shift Work Sleep Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cephalon (Industry)
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C10953/3023/ES/MN
Record Dates: First submitted 2004-02-23; First posted 2004-02-25 (Estimated); Results first posted 2010-02-22 (Estimated); Last update posted 2013-07-19 (Estimated); Status verified 2013-07

CONDITIONS: Narcolepsy; Sleep Apnea, Obstructive; Sleep Apnea Syndromes; Shift-Work Sleep Disorder
Keywords: Excessive Sleepiness; Narcolepsy; Cataplexy; Sleep Attacks; Obstructive Sleep Apnea; Obstructive Sleep Hypopnea; nCPAP; Chronic Shift Work Sleep Disorder; Chronic SWSD; Circadian Rhythm Disorder; Shift Worker; Cepahlon; Cephalon, Inc; Nuvigil
MeSH Terms: conditions — Narcolepsy; Sleep Apnea, Obstructive; Sleep Apnea Syndromes; Sleep Disorders, Circadian Rhythm; Disorders of Excessive Somnolence; Cataplexy; Chronobiology Disorders | interventions — Modafinil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: CEP-10953 (Armodafinil) — Armodafinil (po) 100 to 250 mg/day up to 12 months

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of Armodafinil (CEP-10953) administered on a flexible-dosage regimen of 100 to 250 mg/day for up to 12 months to patients with excessive sleepiness associated with a current diagnosis of narcolepsy, obstructive sleep apnea/hypopnea syndrome (OSAHS)(regular users of nasal continuous positive airway pressure [nCPAP] therapy), or chronic shift work sleep disorder (SWSD).

ELIGIBILITY:
Inclusion Criteria:

Patients are included in the study if all of the following criteria are met:

1. Written informed consent is obtained.
2. Men and women (outpatients) of any ethnic origin, between 18 and 65 years of age (inclusive) are eligible.
3. The patient has a complaint of excessive sleepiness associated with a current diagnosis of:

   * Narcolepsy-Diagnosis made on the basis of International Classification of Sleep Disorders (ICSD) (American Sleep Disorders Association 2000) criteria.
   * OSAHS-Diagnosis made on the basis of ICSD criteria. Furthermore, patients with OSAHS must meet the following nCPAP therapy requirements:

     * Previous adequate education and intervention efforts to encourage nCPAP therapy use must be documented.
     * A patient's nCPAP therapy regimen must be stable for at least 4 weeks.
     * nCPAP therapy is effective, in the opinion of the investigator.
     * Evidence of regular nCPAP usage must be shown during a 2 week evaluation period (ie, nCPAP therapy usage of at least 4 hours/night on at least 70% of the nights).
   * Chronic SWSD-Diagnosis made on the basis of at least minimum ICSD criteria. Furthermore, patients with chronic SWSD must have had excessive sleepiness during night shifts for at least 3 months, work a minimum of 3 night shifts per month that include at least 6 hours between 2200 and 0800 and are no longer than 12 hours in duration, and plan to continue to work night shifts throughout the study.
4. The patient has a Clinical Global Impression of Severity of Disease (CGI-S) rating of 4 or more. (For patients with OSAHS, the CGI-S scale will be administered after nCPAP effectiveness and regular usage is established. For patients with narcolepsy or OSAHS, CGI-S will be evaluated to assess general clinical condition. For patients with SWSD, CGI-S will be evaluated to assess sleepiness during the night shift including the commute to and from work.)
5. The patient is in good health as determined by a medical and psychiatric history, medical examination, electrocardiogram (ECG), serum chemistry and hematology. Women must be surgically sterile, 2 years postmenopausal, or if of childbearing potential, must use a medically accepted method of birth control (ie, barrier method with spermicide, steroidal contraceptive [oral, implanted, and Depo-Provera contraceptives must be used in conjunction with a barrier method], or intrauterine device [IUD]).
6. The patient may have been prescribed PROVIGIL or stimulant therapy to treat the sleep disorder; however, they must have undergone a washout period of at least 7 days prior to screening assessments.
7. The patient must be willing and able to comply with study restrictions and to attend regularly scheduled clinic visits as specified in this protocol.

Exclusion Criteria:

Patients are excluded from participating in this study if 1 or more of the following criteria are met:

1. have any clinically significant, uncontrolled medical conditions (treated or untreated)
2. have a probable diagnosis of a current sleep disorder other than the primary diagnosis of narcolepsy, OSAHS, or chronic SWSD
3. consume caffeine including coffee, tea and/or other caffeine containing beverages or food averaging more than 600 mg of caffeine or more than 8 cups of coffee per day
4. used any prescription drugs disallowed by the protocol or clinically significant use of over-the-counter (OTC) drugs within 7 days before the baseline visit
5. have a history of alcohol, narcotic, or any other drug abuse as defined by the Diagnostic and Statistical Manual of the American Psychiatric Association, 4th Edition (DSM IV)
6. have a positive UDS at the screening visit
7. have a clinically significant deviation from normal in the physical examination
8. are pregnant or lactating. Any woman becoming pregnant during the study will be withdrawn from the study
9. have used an investigational drug within 1 month before the screening visit
10. have any disorder that may interfere with drug absorption, distribution, metabolism, or excretion (including gastrointestinal surgery)
11. have a known clinically significant drug sensitivity to stimulants

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Actual)
Dates: Start 2004-01; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (50):
- United States (41):
  - Pivotal Research Centers, Peoria, Arizona
  - Central Phoenix Medical Clinic, LLC, Phoenix, Arizona
  - Radiant Research - Tucson, Tucson, Arizona
  - Central Arkansas Research, Hot Springs, Arkansas
  - Arkansas Center for Sleep Medicine, Little Rock, Arkansas
  - Bay Area Research Institute, Lafayette, California
  - Pharmacology Research Institute, Los Alamitos, California
  - Neuro-Therapeutics Inc., Pasadena, California
  - Anderson Clinical Research, Redlands, California
  - Synergy Clinical Research Center, San Diego, California
  - BMR HealthQuest Clinical Trials, San Diego, California
  - Rocky Mountain Center for Clinical Research, Wheat Ridge, Colorado
  - Therafirst Medical Centers, Fort Lauderdale, Florida
  - Precision Research, Hallandale, Florida
  - Renstar Medical Research, Ocala, Florida
  - Clinical Research Group of St. Petersburg, St. Petersburg, Florida
  - Radiant Research, Boise, Boise, Idaho
  - Herron Medical Center, Ltd., Chicago, Illinois
  - Radiant Research, Chicago, Chicago, Illinois
  - Radiant Research Alexian Brothers, Elk Grove Village, Illinois
  - Henry W. Lahmeyer, MD and Associates, Northfield, Illinois
  - Vince and Associates Clinical Research, Overland Park, Kansas
  - NeuroTrials Research of New Orleans, LLC, Metairie, Louisiana
  - Marc Raphaelson, MD, PA, Frederick, Maryland
  - Michigan Head-Pain Neurological Institute, Ann Arbor, Michigan
  - Somnos Laboratories, Inc, Lincoln, Nebraska
  - Clinical Research Center of Nevada, Las Vegas, Nevada
  - CNS Research Institute, PC, Clementon, New Jersey
  - Long Island Clinical Research Associates, LLP, Great Neck, New York
  - North Shore University Hospital, Manhasset, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - North Coast Clinical Trials, Inc, Beachwood, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Clinical Research Studies, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital Hospital, Allentown, Pennsylvania
  - Center for Sleep Disorders, Inc., Pottstown, Pennsylvania
  - SleepMed of South Carolina, Columbia, South Carolina
  - Radiant Research, San Antonio, San Antonio, Texas
  - Radiant Research, Salt Lake City, Utah
  - Northwest Clinical Research Center, Bellevue, Washington
- Russia (9):
  - Institute of Pulmonology, Moscow
  - Moscow City Somnological Center, Moscow
  - City Clinical Hospital No. 83, Moscow
  - United Hospital and Out-patient Clinic of Presidential Medical Center of Russian Federation, Moscow
  - City Clinical Hospital No. 81, Moscow
  - Center of Rehabilitation of Presidential Medical Center, Moscow
  - Medical Sanitary Unit No. 122 of Saint-Petersburg, Saint Petersburg
  - Cardioclinic, Saint Petersburg
  - Clinic of Neurology and Neurosurgery of Saint Petersburg, Saint Petersburg

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 41 centers (US 34, Russia 7). First patient enrolled: 30 January 2004/ Last patient last visit: 19 July 2006
Pre-assignment Details: 5 male participants withdrew after enrollment but prior to receiving study drug (1 withdrew consent, 3 were lost to follow-up, and 1 was noncompliant). These 5 patients are in the participant flow, but not in the safety data set since they did not receive study drug.
Groups:
- Armodafinil 100 to 250 mg/Day: Participants with narcolepsy or Obstructive Sleep Apnea/Hypopnea Syndrome (OSAHS): armodafinil once daily in the morning. Participants with chronic Shift Work Sleep Disorder (SWSD): armodafinil 100-250 mg once daily only on nights worked
Period: Overall Study
Arm/Group | Armodafinil 100 to 250 mg/Day
Started | 328
Completed | 151
Not Completed | 177
Not completed — Adverse Event | 43
Not completed — Lack of Efficacy | 15
Not completed — Lost to Follow-up | 41
Not completed — Physician Decision | 9
Not completed — Protocol Violation | 3
Not completed — Withdrawal by Subject | 33
Not completed — Miscellaneous | 33

BASELINE CHARACTERISTICS:
Arm/Group | Armodafinil 100 to 250 mg/Day
Number analyzed (Participants) | 328
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 326
  >=65 years | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 45.2 (11.27)
Gender [Number; unit: participants] — 5 male participants withdrew after enrollment but prior to receiving study drug (1 withdrew consent, 3 were lost to follow-up, and 1 was noncompliant)
  participants
    Female | 111
    Male | 212
Region of Enrollment [Number; unit: participants]
  United States | 267
  Russian Federation | 61

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability as Measured by Number of Participants With Adverse Events
Description: Serious and Non-serious Adverse Events (SAEs). Serious adverse event is any adverse event occurring at any dose that results in any of the following outcomes: death, life-threatening, inpatient hospitalization, persistent or significant disability, congenital anomaly, or an important medical event. An adverse event that does not meet any of the criteria for seriousness listed previously will be regarded as a nonserious adverse event.
Time Frame: Screening/Baseline and months 1, 3, 6, 9, and 12 and every 3 months thereafter
Population: Safety Analysis set of 323 total patients: 5 participants withdrew after enrollment but prior to receiving study drug (1 withdrew consent, 3 were lost to follow-up, and 1 was noncompliant)
Measure: Number; unit: Participants
Arm/Group | Armodafinil 100 to 250 mg/Day
Number analyzed (Participants) | 323
Participants | 323

ADVERSE EVENTS:
Arm/Group | Armodafinil 100 to 250 mg/Day
Serious Adverse Events (participants affected / at risk) | 12/323
Other Adverse Events (participants affected / at risk) | 177/323
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Armodafinil 100 to 250 mg/Day (N=323)
Myocardial infarction (Cardiac disorders) | 1
Tachycardia paroxysmal (Cardiac disorders) | 1
Abdominal haematoma (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 2
Non-cardiac chest pain (General disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Multiple sclerosis (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Menometrorrhagia (Reproductive system and breast disorders) | 1
Chronic obstructive airways disease exacerbated (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Haematoma (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Armodafinil 100 to 250 mg/Day (N=323)
Nausea (Gastrointestinal disorders) | 27
Upper respiratory tract infection (Infections and infestations) | 33
Nasopharyngitis (Infections and infestations) | 18
Sinusitis (Infections and infestations) | 18
Headache (Nervous system disorders) | 55
Dizziness (Nervous system disorders) | 27
Insomnia (Psychiatric disorders) | 46
Anxiety (Psychiatric disorders) | 21
Hypertension (Vascular disorders) | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days